CLINICAL TRIAL: NCT03139695
Title: High Resolution Ultrasound of Intercostal Muscle and Diaphragm as a Biomarker of Respiratory Muscle Function in Patients on Mechanical Ventilation
Brief Title: Using Ultrasound to Study Respiratory Muscle Function in Critically Ill Patients
Status: Completed | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00022412
Record Dates: First submitted 2017-04-19; First posted 2017-05-04 (Actual); Last update posted 2017-11-08 (Actual); Status verified 2017-05

CONDITIONS: Injury of Diaphragm; Mechanical Ventilation Complication; Critical Illness
MeSH Terms: conditions — Critical Illness | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Critically ill patients: High resolution ultrasound of the diaphragm and intercostal muscle
  Interventions: Diagnostic Test: Ultrasound

INTERVENTIONS:
Diagnostic Test: Ultrasound — High resolution Ultrasound of the Diaphragm and Intercostal muscles

SUMMARY:
Mechanical ventilation can be life saving strategy for patients with respiratory failure due to a variety of reasons. Once the underlying illness has resolved, intensive care doctors have to take a decision on when the patient is safe to get off the ventilator or be extubated. They use clinical assessment of the patient's ability to breathe spontaneously and make use of some breathing parameters to make the judgment. Most of the time, a patient can come off the ventilator and do well, but sometimes muscle weakness from sickness can affect the patient's ability to breathe adequately once ventilator support is discontinued. If that occurs, the patient may have to be put back on the ventilator and the physician will suggest some changes to help muscles get stronger. A simple, non-invasive test that can assess respiratory muscle state before taking patients off the ventilator to see if their muscles look healthy can help distinguish which patients may not be ready to be extubated. There are currently several tests available to assess muscle strength, in particular muscles that help in breathing like the intercostal muscles and diaphragm. The study will test the use of Ultrasonography (Ultrasound) as a non-invasive test to assess the muscles of respiration. This test will also help the investigators test physical therapies and interventions of mechanical ventilation that can help patients strengthen the muscles while waiting for extubation.

DETAILED DESCRIPTION:
This is a prospective observational study designed to assess serial changes in quantitative respiratory parameters in patients on different modes of MV e.g. synchronized intermittent mandatory ventilation, controlled mechanical ventilation and pressure support ventilation. This strategy will compare serial changes in diaphragm muscle parameters in ventilator strategies that provide different level of spontaneous respiratory effort and targets for MV. The study will be carried out at Wake Forest Baptist Medical Center. The protocol has been approved by the Institutional Review Board. All adult (>18 years) patients admitted to an ICU will be screened. Written informed consent will be obtained from each patient or their surrogate.

Daily ultrasound studies will be done on the diaphragm muscle. The first study will be conducted within 48 hours of ICU admission. Serial exams will be repeated daily until the patients are extubated or transferred out of the ICU. A maximum of 7 ultrasound studies will be performed since the focus is to demonstrate the utility of early serial changes in measurable parameters on ultrasound. Images will be acquired on both sides during quiet breathing with the patient's arms relaxed by the side in a neutral position while lying with the head of bed at 30 degrees. Most ICU patients are in this position. Diaphragm muscle image at end expiration on each side will be acquired in B mode with a 6-13 MHz transducer in the mid axillary line using the intercostal approach. Diaphragm excursion will be measured bilaterally through anterior subcostal approach in the M mode through a 2-5 MHz transducer. Images will be acquired in accordance with the guidelines set forth in the AANEM position statement. Each ultrasound examination will be done at a time when it does not interfere with concurrent ongoing nursing & medical care.

To determine the effect of the serial changes that occur in respiratory muscle thickness and echodensity on MV, linear regression models will be applied. The distribution of the outcome variables and the need for any transformation to approximate normality will be checked. The outcome variables are serial changes between first and last visit diaphragm muscle thickness and echodensity. The covariate of interest is the mode of MV. The confounding variables are neurological disease, acute lung injury, cumulative fluid balance, age, BMI, history of smoking, duration between the first and last ultrasound examination and the nutritional status (albumin, cumulative calorie intake and type of tube feeds). Since serial changes are the outcome variables, besides the potential confounders, baseline outcome measures will be also adjusted in the regression models. Model selection approaches will be used to select the confounding variables adjusted in the models. Furthermore, to consider the changes across different ultrasound visits, first the individual trajectories of the outcome variables will be displayed graphically. Then, the mixed effects model will be used to examine the associations. This model can handle repeated measures over time by modeling the covariance structure. The covariates will be the same as described previously for the linear regression model. Logistic regression models will then be used to determine if the serial changes in diaphragm muscle thickness and echodensity predict the total number of days on MV, success at SBTs and successful extubation.

Diaphragm ultrasound is a promising new method for evaluating the diaphragm during MV. The investigators feel that the study proposal is extremely relevant in its ability to explore a novel approach to assess the risk of extubation failure, very early on, in the course of MV based on change in muscle echotexture using a noninvasive bedside tool. The investigators propose that changes in diaphragm configuration associated with MV correlate to clinical outcomes as measured by days on MV and extubation failure. The early serial changes detected by ultrasound suggest a potential benefit of proactive early therapies designed to preserve respiratory muscle architecture to reduce days on MV and prevent extubation failure. The investigators further hypothesize that different ventilator modes may affect these changes differentially and these changes might be prevented by titrating ventilatory support to maintain normal levels of respiratory effort. If spontaneously breathing patients and patients on low level of ventilatory support show differential changes on diaphragm muscle parameters compared to patients on controlled modes and higher ventilatory support, clinical protocols might need to emphasize alternate strategies that focus on "muscle protective" or "muscle restorative" ventilation. Ultrasound can also be used to develop clinical paradigms that involve inspiratory muscle training in helping patients who have failed extubation in getting liberated from MV.

The goals are to use the pilot data generated through this grant to power and design a randomized controlled trial of a "muscle protective" or "muscle restorative" ventilation strategy and assess its effectiveness in reducing days on MV and extubation failure compared to current medical practice. This team approach will involve a novel collaboration of key members with expertise in muscle ultrasound, mechanical ventilation, mechanisms of muscle wasting related to acute lung injury and physiological effects of exercise on respiratory muscle hence representing critical input into developing clinical strategies to assess and reduce the burden of extubation failure. The investigators believe this approach is innovative in aiming to use a non-invasive bedside clinical tool to develop "muscle protective" and "muscle restorative" ventilator strategies with a focus on early respiratory rehabilitation in critically ill patients on MV.

ELIGIBILITY:
Inclusion Criteria

* Patients will be included if first ultrasound measurement can be performed within 48 hours of ICU admission and informed consent can be obtained from patient or designated health care representative.
* Adult patients (≥ 18 years of age) in any intensive care unit.
* Patients who are expected to have the need for prolonged mechanical ventilation (treating physician's assessments that patient will likely need mechanical ventilation for >48 hours; 2 days) and have been on mechanical ventilation for <48 hours at the time of enrollment.

Exclusion Criteria

* Patients in any ICU who is expected to be on mechanical ventilation for <48 hours based on treating physicians judgment.
* Patients that were on MV for more than 48 hours prior to transfer to the ICU.
* Patients who are expected to be extubated, transferred out of the ICU or discharged from the intensive care unit in the next 48 hours based on treating physicians judgment.
* Patients who are transitioning to palliative care or expected to die in the next 48 hours based on treating physicians judgment.
* Any patient where access to chest to study intercostal muscle and diaphragm is limited due to skin /subcutaneous lesions.
* Patients with a history of or current chest tubes, chest trauma or anterior rib fractures.
* Patients with a history of prior MV >48 hours or prior history of tracheostomy.
* Patients with a history of chest or abdominal surgery.
* Patients that have a tracheotomy or require non-standard modes of ventilation including airway pressure release ventilation or high frequency oscillatory ventilation.
* Patients with physician orders for positioning of the patient is different from head of the bed at 30 degree. E.g. patients with recent lumbar spinal surgery are laid flat to reduce spinal fluid pressure in lumbar area.
* Patients with a known allergy to ultrasound gel
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients (≥ 18 years of age) in intensive care unit
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2012-11; Primary Completion 2016-07-01 (Actual); Study Completion 2016-07-01 (Actual)

PRIMARY OUTCOMES:
Change from Baseline of thickening fraction of diaphragm muscle | 7 days
  Muscle thickness will be measured at end inspiration and end expiration images of diaphragm to ascertain the thickening fraction of the diaphragm. Progression of muscle thickening fraction during mechanical ventilation will be assessed.

SECONDARY OUTCOMES:
Change from Baseline of Echodensity of diaphragm muscle | 7 days
  Muscle echodensity will be ascertained using Gray scale histogram analysis ( using Image J ) on images of diaphragm to ascertain the echodensity of the diaphragm. Progression of muscle echodensity during mechanical ventilation will be assessed.
Change from Baseline of thickness of intercostal muscle | 7 days
  Muscle thickness will be measured on images of intercostal muscles. Progression of muscle thickenness during mechanical ventilation will be assessed.
Change from Baseline of Echodensity of intercostal muscle | 7 days
  Muscle echodensity will be ascertained using Gray scale histogram analysis ( using Image J ) on images of intercostal muscle to ascertain the echodensity of intercostal muscle. Progression of muscle echodensity during mechanical ventilation will be assessed.
Duration of mechanical ventilation | Through study completion, expected less than 6 months
  Results will be analyzed initially using descriptive statistics. Comparison between groups will be done using chi square tests for proportions, and t-tests or ANOVA procedures for continuous variables. Regression analysis will be performed to identify independent outcome predictors. Other inferential statistical analysis will be conducted as appropriate.
Success / failure at spontaneous breathing trials | Through study completion, expected less than 6 months
  Results will be analyzed initially using descriptive statistics. Comparison between groups will be done using chi square tests for proportions, and t-tests or ANOVA procedures for continuous variables. Regression analysis will be performed to identify independent outcome predictors. Other inferential statistical analysis will be conducted as appropriate.
Success at first extubation | Through study completion, expected less than 6 months
  Results will be analyzed initially using descriptive statistics. Comparison between groups will be done using chi square tests for proportions, and t-tests or ANOVA procedures for continuous variables. Regression analysis will be performed to identify independent outcome predictors. Other inferential statistical analysis will be conducted as appropriate.
Overall duration of mechanical ventilation during hospital stay | Through study completion, expected less than 6 months
  Results will be analyzed initially using descriptive statistics. Comparison between groups will be done using chi square tests for proportions, and t-tests or ANOVA procedures for continuous variables. Regression analysis will be performed to identify independent outcome predictors. Other inferential statistical analysis will be conducted as appropriate.
Total length of ICU stay | Through Study completion, expected less than 6 months
  Results will be analyzed initially using descriptive statistics. Comparison between groups will be done using chi square tests for proportions, and t-tests or ANOVA procedures for continuous variables. Regression analysis will be performed to identify independent outcome predictors. Other inferential statistical analysis will be conducted as appropriate.

CONTACTS AND LOCATIONS:
Overall Officials: Aarti Sarwal, MD, Principal Investigator — Wake Forest UBMC
Locations (1):
- Wake Forest Univesity Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sarwal A, Liu A, Cartwright MS, Dhar S, Morris PE. Sonography for Assessing Dynamic Diaphragm Dysfunction in Acute Respiratory Distress. J Ultrasound Med. 2015 Sep;34(9):1701-6. doi: 10.7863/ultra.15.14.10047. Epub 2015 Aug 17. No abstract available. PMID 26283757
- [Background] Parry SM, El-Ansary D, Cartwright MS, Sarwal A, Berney S, Koopman R, Annoni R, Puthucheary Z, Gordon IR, Morris PE, Denehy L. Ultrasonography in the intensive care setting can be used to detect changes in the quality and quantity of muscle and is related to muscle strength and function. J Crit Care. 2015 Oct;30(5):1151.e9-14. doi: 10.1016/j.jcrc.2015.05.024. Epub 2015 Jun 3. PMID 26211979
- [Background] Sarwal A, Parry SM, Berry MJ, Hsu FC, Lewis MT, Justus NW, Morris PE, Denehy L, Berney S, Dhar S, Cartwright MS. Interobserver Reliability of Quantitative Muscle Sonographic Analysis in the Critically Ill Population. J Ultrasound Med. 2015 Jul;34(7):1191-200. doi: 10.7863/ultra.34.7.1191. PMID 26112621
- [Background] Sarwal A, Cartwright MS, Walker FO, Mitchell E, Buj-Bello A, Beggs AH, Childers MK. Ultrasound assessment of the diaphragm: Preliminary study of a canine model of X-linked myotubular myopathy. Muscle Nerve. 2014 Oct;50(4):607-9. doi: 10.1002/mus.24294. Epub 2014 Aug 30. PMID 24861988
- [Background] Sarwal A, Cartwright MS, Mitchell E, Williams K, Walker FO, Childers MK. Guiding intramuscular diaphragm injections using real-time ultrasound and electromyography. Muscle Nerve. 2015 Feb;51(2):287-9. doi: 10.1002/mus.24493. PMID 25354257
- [Background] Sarwal A, Walker FO, Cartwright MS. Neuromuscular ultrasound for evaluation of the diaphragm. Muscle Nerve. 2013 Mar;47(3):319-29. doi: 10.1002/mus.23671. Epub 2013 Feb 4. PMID 23382111
- [Background] Cartwright MS, Kwayisi G, Griffin LP, Sarwal A, Walker FO, Harris JM, Berry MJ, Chahal PS, Morris PE. Quantitative neuromuscular ultrasound in the intensive care unit. Muscle Nerve. 2013 Feb;47(2):255-9. doi: 10.1002/mus.23525. Epub 2012 Oct 5. PMID 23041986
- [Background] Morris PE, Berry MJ, Files DC, Thompson JC, Hauser J, Flores L, Dhar S, Chmelo E, Lovato J, Case LD, Bakhru RN, Sarwal A, Parry SM, Campbell P, Mote A, Winkelman C, Hite RD, Nicklas B, Chatterjee A, Young MP. Standardized Rehabilitation and Hospital Length of Stay Among Patients With Acute Respiratory Failure: A Randomized Clinical Trial. JAMA. 2016 Jun 28;315(24):2694-702. doi: 10.1001/jama.2016.7201. PMID 27367766